CLINICAL TRIAL: NCT02607449
Title: Randomized, Placebo-controlled Study of Safety and Therapeutic Efficacy of the Drug FS-1 in the Oral Dosage Form in Drug-resistant Pulmonary Tuberculosis
Brief Title: FS-1 Drug for Treatment of Multiple Drug-resistant Tuberculosis
Acronym: FS-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scientific Center for Anti-infectious Drugs, Kazakhstan (Industry)
Collaborators: Phthisiopulmonology Center of Almaty, Kazakhstan (Unknown); National Scientific Center of Phthisiopulmonology, Kazakhstan (Unknown); Karaganda Medical University (Other); West Kazakhstan Marat Ospanov Medical University, Aktobe, Kazakhstan (Unknown); Semey State Medical University (Other); National Center of Phthisiatry, Bishkek, Kyrgyzstan (Other); Invivo laboratory, Kazakhstan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TP-004 V 5.1
Record Dates: First submitted 2015-11-11; First posted 2015-11-18 (Estimated); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Tuberculosis, MDR
Keywords: Tuberculosis; Multi-drug resistant TB; TB treatment
MeSH Terms: conditions — Tuberculosis, Multidrug-Resistant; Tuberculosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): Standard TB treatment+ treatment regiment with FS-1 drug. Study drug was given to the patients orally once per day in dose of 2.5 mg/kg along with other prescribed TB drugs.
  Interventions: Drug: FS-1
- B (Placebo Comparator): Standard TB treatment + treatment regiment with a placebo. Instead of study drug the placebo was given to the patients orally once per day along with other prescribed TB drugs (in quntity equal to study drug).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FS-1 — FS-1 is a liquid solution for internal intake and has antimicrobial and antibacterial activities.
  Arms: A
Drug: Placebo — Placebo without any active pharmaceutical ingredients
  Arms: B

SUMMARY:
Drug-resistant tuberculosis is becoming a major problem for the whole humanity, and development of new Anti-TB drugs is of great importance. Since Kazakhstan is a country with the high burden of tuberculosis, the Government of the Republic of Kazakhstan has founded initiative on the development of new Anti-TB drug to treat drug-resistant forms of this infectious disease. JSC "Scientific Center for Anti-infectious Drugs" has developed original drug FS-1 for the treatment of multidrug resistant tuberculosis (MDR-TB).

DETAILED DESCRIPTION:
Phase 3 clinical study of FS-1 drug is a randomized, interventional, multicenter, placebo-controlled (add-on), double-blind and two arms trial.

The study consists of two following phases: treatment phase - 6 months and follow-up phase 12 months. It is planned to recruit 480 patients with verified MDR-TB diagnosis.

All data will be compiled in an Electronic Data Capture System with further statistical analysis according to approved Statistical Analytical Plan.

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from a multidrug-resistant form of pulmonary tuberculosis which is defined by:

  * MDR Tuberculosis confirmed by microbiology test at screening.
  * resistance to isoniazid and rifampicin demonstrated by drug susceptibility test
  * susceptiblity of TB bacteria to fluoroquinolones and aminoglycoside/capreomycin
* all ethnicities, intellectually capable of understanding their own condition and the requirements of the study protocol
* Willing to freely and voluntarily give signed informed consent
* Willing and capable to comply with all requirements of the protocol

Exclusion Criteria:

* Pregnancy and breast-feeding;
* Patients with decompensated concomitant diseases (cardiovascular, renal, hepatic failure) that may affect the conduct of the study;
* Severe mental disorders;
* Allergy to iodine-containing drugs, hypersensitivity to iodine;
* Intolerance to second-line drugs;
* Epidermomycosis
* Socially maladjusted patients suffering from alcoholism and drug addiction;
* Hypothyroidism;
* Hashimoto's thyroiditis;
* TB treatment for more than two months before the start of the study;
* Not willing to adhere to TB therapy;

Exclusion Criteria during the study:

* at the discretion of the researcher, if the continuation of the study is harmful to the patient;
* side effects related with the study drug
* patient's decision to stop participation in study
* appearance of any exclusion criteria during study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2020-08 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Time to persistently negative sputum cultures | 18 months
  Time from the start of treatment with study drug to the first negative M. tuberculosis sputum culture on solid medium followed by 4 consecutive negative results with an interval of at least 30 days. Measured in months. Estimated population: randomized subjects who took at least 70% of planned study drug doses; having a positive bacterial culture M. tuberculosis at the baseline; who missed less than 2 consecutive visits or less than 14 consecutive days of study drug treatment (modified ITT analysis).
Proportion of Patients with persistently negative sputum cultures (SCC) | 12 months
  Sputum culture conversion (SCC) is a persistently negative result of the sputum culture at one year from the patients who had sputum samples positive for growth of M. tuberculosis at baseline and not followed by any positive culture until the end of the trial. SCC corresponds to the outcome "cured" if at least 5 negative bacteriological cultures is recorded (on solid medium) during 12 months with an interval of at least 30 days.

SECONDARY OUTCOMES:
The proportion of subjects with relapse of tuberculosis | 12 months
  Relapse is defined when patient received full study drug treatment course (6 months) and bacteriological culture become again positive after 5 negative bacteriological cultures (on solid medium) during 12 months with an interval of at least 30 days.
Patients body weight dynamics for the period of 18 months. | 18 months
  Comparison of subjects' weight, using as the baseline subjects' weight before the start of the treatment with the subjects' weight during the treatment cycle with the study drug (6 months) and during 12 months of follow-up period.
The median time to occurrence of negative sputum microscopy result | 18 months
  The average time between positive and negative sputum smear microscopy results during the treatment.
The time when TB clinical symptoms not observed | 18 months
  Assessment of period between TB clinical symptoms and their disappearance. Observed of TB clinical symptoms are as follows: chest pain, difficulties to breath, cough, sputum, intoxication symptoms.
Dynamics of the tuberculosis process based on subjects chest x-ray diagnosis. | 18 months
  The positive dynamics of the subject X-ray picture of the tuberculous process is characterized by the closure of TB caused cavities, a decrease of lung infiltration, nodular lesions, pleural effusion and lymphadenopathy.
The incidence and severity of Adverse Events, Serious Adverse Events and drug related Adverse Drug Reactions | 18 months
  Assessment of Adverse Events and Drug Reactions during the study (6 months of treatment and 12 months of follow-up period).
  Adverse event (AE) is any untoward medical occurrence in subject administered the study drug and that does not necessarily have a causal relationship with this treatment. AE is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a study drug, whether or not related to the study drug.
  Serious Adverse Event is any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect.
  Adverse drug reaction - all noxious and unintended responses to the study drug, when a causal relationship between the study drug and an adverse event is at least a reasonable possibility.
Assessment of the study drug effect on thyroid gland function | 18 months
  Assessment of thyroid hormones and antibodies in the blood (free triiodothyronine (FT3), free thyroxine (FT4), total thyroxine (TT4),total triiodothyronine (TT3),thyroid stimulating hormone (TSH), antibodies to thyroglobulin and thyroid peroxidase), and results of ultrasound of the thyroid gland before treatment, during treatment (6 months) and during the follow-up period (12 months).

CONTACTS AND LOCATIONS:
Overall Officials: Amirkan A Azembayev, Cond.Phar.Sc., Study Director — JSC "Scientific Center for Anti-infectious Drugs"
Locations (6):
- Kazakhstan (5):
  - Semey Medical University, Semey, East Kazakhstan
  - West Kazakhstan Marat Ospanov Medical University, Aktobe, West Kazakhstan
  - National scientific center of phthisiopulmonology Ministry of health of the Republic of Kazakhstan, Almaty
  - Center of Phthisiopulmonology of the Public Health Administration of Almaty, Almaty
  - Karaganda Medical University, Karaganda
- National Center of Phthisiatry, Bishkek, Kyrgyzstan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Genomic Insight into Mechanisms of Reversion of Antibiotic Resistance in Multi-Drug Resistant Mycobacterium Tuberculosis Induced by FS-1 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC5420568/
- See also: Complete genome sequence of the multi-drug resistant clinical isolate Mycobacterium tuberculosis 187.0 used to study an effect of drug susceptibility reversion by drug FS-1 — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4645197/
- See also: Constraints of Drug Resistance - Prospects for Pharmacological Reversion of Susceptibility to Antibiotics — https://pdfs.semanticscholar.org/aa99/f23a56e4984ce275274125c48c23ee3cba10.pdf?_ga=2.196299177.40052518.1562695622-2113992793.1562695622
- See also: The effect of the Kazakhstan drug FS-1 on the outcome of multidrug-resistant pulmonary tuberculosis in complex anti-tuberculosis therapy — http://sbook.ru/vrasp/contents/va15711sd.pdf
- See also: Anti-tuberculosis activity of new drug FS-1 — http://sibac.info/conf/med/xliv/42595